CLINICAL TRIAL: NCT05135130
Title: A Retrospective Record-review Study in Patients Who Had Participated in the ON101CLCT02 Diabetic Foot Ulcer Trial
Brief Title: Retrospective Record-review Study in Patients Who Had Diabetic Foot Ulcer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Oneness Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: ON101CLOS01
Record Dates: First submitted 2021-11-16; First posted 2021-11-26 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ON101 Cream: Patients Who Had Participated in the ON101CLCT02 Diabetic Foot Ulcer Trial and assigned to ON101 Cream arm
  Interventions: Drug: ON101 Cream
- Aquacel® Hydrofiber® dressing: Patients Who Had Participated in the ON101CLCT02 Diabetic Foot Ulcer Trial and assigned to Aquacel® Hydrofiber® dressing arm

INTERVENTIONS:
Drug: ON101 Cream — Not applicable in this retrospective study
  Groups: ON101 Cream

SUMMARY:
The purpose of the study is to evaluate the medical cost of illness for DFUs on the patients who had used ON101 or Aquacel® in the ON101CLCT02 trial.

ELIGIBILITY:
No additional inclusion or exclusion criteria will be applied.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The ON101CLCT02 trial enrolled 236 subjects and was conducted in Taiwan, China, and USA. The target population of this study consists of the Taiwanese DFU patients who had completed or early withdrawn from the ON101CLCT02 trial.
Sampling Method: Non-Probability Sample
Enrollment: 176 (Estimated)
Dates: Start 2021-10-04 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Demographic characteristics | Up to two years after the patient had completed or early withdrawn from the ON101CLCT02 trial
Wound characteristics of DFUs (classification and proportion) | Up to two years after the patient had completed or early withdrawn from the ON101CLCT02 trial
Proportion of DFU recurrence after completing or withdrawing from the ON101CLCT02 trial | Up to two years after the patient had completed or early withdrawn from the ON101CLCT02 trial
Medical costs due to DFUs | Up to two years after the patient had completed or early withdrawn from the ON101CLCT02 trial
Proportion of wound infection, gangrene, and amputation | Up to two years after the patient had completed or early withdrawn from the ON101CLCT02 trial
Frequency of wound infection, gangrene, and amputation | Up to two years after the patient had completed or early withdrawn from the ON101CLCT02 trial

CONTACTS AND LOCATIONS:
Overall Officials: Shyi-Gen Chen, MD, Study Director — Oneness Biotech Co., Ltd.
Locations (1):
- China Medical University Hospital, Taichung, Taiwan